CLINICAL TRIAL: NCT05882110
Title: Amplification of Autologous Epidermal Cells to Repair Large Area Deep Wounds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yicheng Ma (Other)
Responsible Party: Sponsor-Investigator, Yicheng Ma, Investigator, First Affiliated Hospital of the Chinese People's Liberation Army Naval Medical University
Organization: First Affiliated Hospital of the Chinese People's Liberation Army Naval Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOAECTRLADW
Record Dates: First submitted 2023-05-02; First posted 2023-05-31 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Autologous Epidermal Cell Transplantation
Keywords: autologous; epidermal cell; transplantation; amplification; deep wounds

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with a body surface wound of 30% TBSA or more and requiring at least 2 weeks to repair (Experimental)
  Interventions: Procedure: Cultured autologous epidermal cell membrane

INTERVENTIONS:
Procedure: Cultured autologous epidermal cell membrane — The cultured autologous epidermal cell membrane is made from the patient's autologous epidermal cells by in vitro rapid expansion and culture technology, which has good biocompatibility, non-toxic, non-teratogenic, can reduce the skin area cut by traditional autologous skin grafting methods, and has high proliferative activity to promote wound repair and regeneration.

SUMMARY:
Autologous epidermal cell transplantation is based on the principle and technology of skin tissue engineering, and is performed by cutting small pieces of autologous skin from patients, isolating and culturing and expanding them, and then transplanting them to the patient's wounds to repair the damage.

DETAILED DESCRIPTION:
Timely wound repair has been a great challenge in the treatment of patients with large deep burns. The current conventional approach is to use autologous skin grafts, such as micro-skin grafts, stamp skin grafts, and mesh skin grafts. Since there is very little normal skin left after large deep burns and the expansion of autologous skin grafts is limited (3-15 times), repeated skin grafting procedures are needed to repair the wound gradually, resulting in a long course of disease, scar growth and contracture, which seriously affects the quality of survival and even endangers life. Especially for patients with very large deep burns, there is an extreme shortage of normal skin sources, so they face the dilemma of having no rice to cook and unable to repair their wounds.

Based on the principle and technology of skin tissue engineering, autologous epidermal cell transplantation can provide sufficient skin source for patients with large deep burns by cutting very small pieces of autologous skin (about 2-10 cm2) and expanding them by 1000-5000 times after 2-3 weeks of in vitro culture. Autologous epidermal cell membranes combined with a large proportion of expanded autologous dermis (e.g. stamp skin, reticular skin) can significantly shorten the interstitial fusion time, improve the survival rate of autologous dermis transplants, and reduce scar growth after wound healing; autologous epidermal cell membranes combined with allogeneic dermis transplants can repair third-degree burn wounds, thus providing a large number of dermis sources for patients with lack of dermis sources, and has become an important treatment tool for saving the lives of patients with large deep burns. It has become an important treatment tool to save the lives of patients with large deep burns.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a body surface trauma of 30% TBSA or more and a wound that requires at least 2 weeks to repair as assessed by the clinician

Exclusion Criteria:

* Patient body surface trauma area less than 30% TBSA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Take rate of cultured epidermal autograft | 4 weeks
  The take rates of CEA(cultured epidermal autograft) were calculated separately for every graft site according to the anatomical regions.
The incidence of serious adverse events | week 52 after applying CEA
  The safety of CEA(cultured epidermal autograft) is evaluated using the incidence of serious adverse events, such as tumorous conditions, allergic reactions, or critical infections.

CONTACTS AND LOCATIONS:
Locations (1):
- Yicheng Ma, Shanghai, Shanghai Municipality, China